CLINICAL TRIAL: NCT04474444
Title: Ambulance Calls for Substance Use and Alcohol in a Pandemic (ASAP): Exploring Attendance at Incidents Involving Substance and/or Alcohol Use During COVID-19 Pandemic
Brief Title: Ambulance Calls for Substance Use and Alcohol in a Pandemic (ASAP)
Acronym: ASAP
Status: Completed | Type: Observational
Sponsor: University of Lincoln (Other)
Responsible Party: Sponsor
Other Study IDs: ASAP01
Record Dates: First submitted 2020-07-12; First posted 2020-07-16 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2020-07

CONDITIONS: Alcohol Use, Unspecified; Substance Use; Intoxication Alcohol; Emergencies; COVID-19 Pandemic; Treatment
MeSH Terms: conditions — Alcohol Drinking; Substance-Related Disorders; Alcoholic Intoxication; Emergencies; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hear and treat: phone call, treatment, not attended
- See and treat: Ambulance crew attended
  Interventions: Other: attendance by ambulance crew

INTERVENTIONS:
Other: attendance by ambulance crew — hear, attendance, convey
  Groups: See and treat

SUMMARY:
The Primary objective is to explore ambulance service attendance at incidents involving alcohol and/or substance use over the period of the pandemic lockdown, and the following months. This will be to determine prevalence and explore factors such as patient gender, age, ethnicity or location. Analysis will examine the calls over the course of the year prior to the lockdown, and then compare this to the period of lockdown and following months.

DETAILED DESCRIPTION:
The Primary objective is to explore ambulance service attendance at incidents involving alcohol and/or substance use over the period of the pandemic lockdown, and the following months. This will be to determine prevalence and explore factors such as patient gender, age, ethnicity or location. Analysis will examine the calls over the course of the year prior to the lockdown, and then compare this to the period of lockdown and following months.

A time series analysis will be conducted to examine the calls over the course of the year prior to the lockdown, and then compare this to the period of lockdown and following months. This will use the 'Interrupted Time Series' (ITS) approach. To explore this regression models will be built that examine the causal models for attendance prior to the pandemic and compared to the lockdown time frame.

A multivariable regression model will be built. Initially a Directed Acyclic Graph (DAG) will allow the identification of confounders and exposures relevant to the model. A logistic regression model will be used to calculate the relative risk of call during lockdown compared to the data prior to lockdown. The model will be fit using p<0.05 as the definition of statistical significance.

Descriptive statistics, trend analysis and predictive analysis will be conducted on the data set to determine trends across time, factors that predict patients requiring ambulance attendance, and factors that predict treatment outcomes. Missing data will be examined for systematic bias, and where found to be missing at random will be excluded from analysis. Where not missing at random, sensitivity analysis will be conducted.

Analysis will examine covariates. Age will be defined as single year continuous variable and examined in categories such as 5-year age groups. Ethnicity will be categorised as groups, such as black, Asian, other minority and mixed ethnic groups will be explored. Census data such as the deprivation, rurality, income, employment, disability and education will look at the decile as defined.

ELIGIBILITY:
Inclusion Criteria:

* Patient of any age
* Patient requested ambulance attendance between 23rd March 2019 and 22nd March 2021
* The patient record is held by East Midlands Ambulance Service
* Patient records that have recorded a clinical impression related to alcohol and substance use will be included in the data set alongside a word search in the free text response box for the following words/phrases: narcotic, spice, mamba, alcohol, substance use, drug use, illicit drug, overdose, intoxication, intoxicated, drunk, high.

Exclusion Criteria:

* The patient record was outside of the indicated date range.
* The patient record is not accessible via EMAS

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All people who ring 999 or 111 in an emergency.
Sampling Method: Non-Probability Sample
Enrollment: 55000 (Actual)
Dates: Start 2019-03-23 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
Attendances for alcohol and drug use | Full data set 23/03/2019 compared to 22/03/2021 to look at interruption (lockdown) in the time series.
  Counts of attendances for alcohol and drug use by the East Midland's Ambulance Service over the time period. This will be a number per day of people attended.

CONTACTS AND LOCATIONS:
Overall Officials: Graham Law, PhD, Principal Investigator — University of Lincoln
Locations (1):
- University of Lincoln, Lincoln, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the IPD